CLINICAL TRIAL: NCT06890689
Title: Effectiveness of Scaling and Root Planing in Deeper Pockets
Status: Active, not recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: Effectiveness of SRP
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Periodontal Disease; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients received SRP at predoctoral clinic
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Retrospective study to evaluate the outcome of scaling and root planing

SUMMARY:
This study will retrospectively evaluate the outcomes of scaling and root planing over a two year time period. The study will focus specifically on the effectiveness of SRP in pockets with an initial pre-treatment pocket probing depth of ≥ 5 mm and ≤ 8 mm. The study will also examine the response to SRP of all initial pocket depths, i.e., those PPD that fall below or above those in the indicated range, to verify the findings of previous studies.

ELIGIBILITY:
Inclusion criteria:

* All patients treated by dental students who have the required data
* 14 or more permanent teeth
* Have at least 2 molars (excluding third molars)

Exclusion Criteria:

* All third molars and second molars next to a partially impacted third molar
* Smokers
* Diabetes
* Immunocompromised patients (HIV/AIDS; chemotherapy; systemic steroid therapy, etc.)
* Pregnancy during treatment or during the follow-up periods
* Diagnosis of Alzheimer's or dementia
* Diagnosis of oral mucous membrane disease (BMMP, Lupus, erosive lichen planus, etc.)
* Patients that have received periodontal surgery following SRP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by dental students at TAMU Collage of Dentistry Predoctoral Clinic
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of SRP (scaling and root planing) in pockets with an initial (baseline) pre-treatment pocket probing depth of ≥ 5 mm and ≤ 8 mm | From January 2020 to January 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University Collage of Dentistry,, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No